CLINICAL TRIAL: NCT02205138
Title: A Pilot Phase 2a, Multicentre, Open, Proof-of-concept Study on the Safety and the Efficacy of Allogeneic Osteoblastic Cells (ALLOB®) Implantation in Lumbar Spinal Fusion
Brief Title: Phase 2a Study on Allogeneic Osteoblastic Cells Implantation in Lumbar Spinal Fusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bone Therapeutics S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLOB-IF1
Record Dates: First submitted 2014-07-30; First posted 2014-07-31 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Degenerative Disc Disease
Keywords: Spinal Fusion; Lumbar Interbody Fusion; Degenerative Disc Disease; Cell Therapy; Bone Graft
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALLOB® cells with ceramic scaffold (Experimental): ALLOB® cells with ceramic scaffold Implantation
  Interventions: Drug: ALLOB® cells with ceramic scaffold

INTERVENTIONS:
Drug: ALLOB® cells with ceramic scaffold — Each patient will undergo a single administration of ALLOB®/ceramic scaffold mix into the lumbar interbody fusion site under anaesthesia

SUMMARY:
Among existing surgical techniques, spinal fusion is considered as the gold standard to treat a broad spectrum of degenerative spine disorders, including spondylolisthesis and scoliosis, with regard to pain reduction and functional improvement. However, pseudarthrosis and failure to relieve low back pain are unfortunately still frequent, irrespective of the type of procedures and grafts used by the surgeon.

The present Phase 2a study aims at demonstrating the safety and efficacy of ALLOB®, a proprietary population of allogeneic osteoblastic cells, in lumbar spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide a written, dated, and signed informed consent prior to any study related procedure, and to understand and comply with study requirements
* Symptomatic degenerative disc disease of the lumbar spine requiring a single level lumbar fusion (L1-S1)
* Unresponsive to non-operative treatment for at least 6 months

Exclusion Criteria:

* Lumbar disc disease requiring treatment at more than one level
* Previous failed fusion at the involved lumbar level
* Local active or latent infection at the involved lumbar level
* Positive serology for hepatitis B, hepatitis C, HIV
* Current or past medical disease that could interfere with the evaluation of the safety and efficacy, as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-10; Primary Completion 2019-02 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Lumbar fusion progression as assessed by CT scan | 12 months
Functional Disability using Oswestry Disability Index | 12 months
Potential occurrence of any AE or SAE, related to the product or to the procedure, using patient open non-directive questionnaire, physical examination and laboratory measurements | 12 months

SECONDARY OUTCOMES:
Pain using a Visual Analogue Scale | 12 months
Global Disease Evaluation using a Visual Analogue Scale | 12 months
Functional Disability using Oswestry Disability Index | 12 months
Lumbar fusion progression as assessed by CT scan | 12 months
Percentage of patients having a rescue surgery | 12 months
Potential occurrence of any AE or SAE related to the product or to the procedure | 36 months

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (8):
  - Investigating site BE01, Brussels
  - Investigating site BE03, Brussels
  - Investigating site BE05, Brussels
  - Investigating site BE02, Charleroi
  - Investigating site BE04, Genk
  - Investigating site BE08, Kortrijk
  - Investigating site BE07, Liège
  - Investigating site BE06, Mons